CLINICAL TRIAL: NCT06021561
Title: Orofacial Pain in Multiple Sclerosis
Status: Withdrawn | Type: Observational
Why Stopped: the principal investigator changed her mind and gave up from the study
Sponsor: Varazdin General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 21062023
Record Dates: First submitted 2023-08-18; First posted 2023-09-01 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis
Keywords: facial pain; craniofacial pain; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Facial Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple sclerosis group: Multiple sclerosis patients registered in Varazdin General Hospital from 1 January 2017 - 31 December 2022
  Interventions: Diagnostic Test: Diagnosis of pain

INTERVENTIONS:
Diagnostic Test: Diagnosis of pain — Pain will be investigated - type, origin, level

SUMMARY:
Although the orofacial pain is not typical symptom of multiple sclerosis, more than 50% of the patients experience some kind of pain. Acute pain usually in form of trigeminal neuralgia, that occurred in 2-3% of patients with multiple sclerosis. Chronic pain occurred in 40-50% of patients and most common forms are headache. Aim of this study is to investigate prevalence and evaluate the form of orofacial pain in patients with multiple sclerosis treated in General hospital Varaždin in period from 01.01. 2017. to 31.12.2022. Results of this investigation will determine better understanding orofacial pain , treatment and impact on everyday life.

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic autoimmune disease with an unknown mechanism of origin. Although pain is not a typical symptom of multiple sclerosis, it occurs in more than 50% of patients and has significant impact on the quality of life of patients. Pain syndromes that patients with multiple sclerosis initially have characteristics of somatic and nociceptive pain, and later neuropathic, including trigeminal neuralgia, headaches, Lhermitte's syndrome.

Pain is also often associated with anxiety and depression, which occurs in almost one third of patients.

Pain therapy in these patients is a challenge for many doctors involved in the treatment. Many patients do not have adequate pain therapy due to the disproportion between the fear of interaction with other drugs and side effects, and on the other hand the treatment of basic diseases with the aim of controlling the immune response.

ELIGIBILITY:
Inclusion Criteria:

* multiple scerosis
* age 18-85 years

Exclusion Criteria:

* records with missing data

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple sclerosis patients aged 18-65 years registered in Varazdin General Hospital from 1 January 2017 to 31 December 2022
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The frequency of orofacial pain in patients with multiple sclerosis | 3 months
  To investigate that, hospital records will be reviewed. Additionally, all of the patients will be approached with the questionnaire investigating the frequency of orofacial pain (expressed in number and proportion of all patients)
The location of orofacial pain in patients with multiple sclerosis | 3 months
  To investigate that, hospital records will be reviewed. Additionally, all of the patients will be approached with the questionnaire investigating the loacation of orofacial pain
The duration of orofacial pain in patients with multiple sclerosis | 3 months
  To investigate that, hospital records will be reviewed. Additionally, all of the patients will be approached with the questionnaire investigating the duration of orofacial pain (in months)

SECONDARY OUTCOMES:
MS therapy's influence to pain | 3 months
  To investigate connection between orofacial pain and multiple sclerosis therapy
MS orofacial pain and the duration of the disease | 3 months
  To investigate the connection between orofacial pain and the duration of the disease
Pain and patients' characteristics | 3 months
  To investigate the pain characteristics in relation to age, sex, form of the disease
Other chronic diseases and orofacial pain | 3 months
  To investigate the influence of other chronic diseases on orofacial pain in patients with multiple sclerosis
Pain and daily functioning | 3 months
  To investigate the impact of pain on the daily functioning of patients with multiple sclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Monika Kocman Panic, MD, Principal Investigator — Varazdin General Hospital, Varazdin, Croatia
Locations (1):
- Varazdin General Hospital, Varaždin, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Putzki N, Pfriem A, Limmroth V, Yaldizli O, Tettenborn B, Diener HC, Katsarava Z. Prevalence of migraine, tension-type headache and trigeminal neuralgia in multiple sclerosis. Eur J Neurol. 2009 Feb;16(2):262-7. doi: 10.1111/j.1468-1331.2008.02406.x. Epub 2008 Dec 9. PMID 19138330
- [Background] Young J, Amatya B, Galea MP, Khan F. Chronic pain in multiple sclerosis: A 10-year longitudinal study. Scand J Pain. 2017 Jul;16:198-203. doi: 10.1016/j.sjpain.2017.04.070. Epub 2017 May 24. PMID 28850402
- [Background] Hirsh AT, Turner AP, Ehde DM, Haselkorn JK. Prevalence and impact of pain in multiple sclerosis: physical and psychologic contributors. Arch Phys Med Rehabil. 2009 Apr;90(4):646-51. doi: 10.1016/j.apmr.2008.10.019. PMID 19345781
- [Background] Di Stefano G, Maarbjerg S, Truini A. Trigeminal neuralgia secondary to multiple sclerosis: from the clinical picture to the treatment options. J Headache Pain. 2019 Feb 19;20(1):20. doi: 10.1186/s10194-019-0969-0. PMID 30782116
- [Background] Kahraman T, Ozdogar AT, Ertekin O, Ozakbas S. Frequency, type, distribution of pain and related factors in persons with multiple sclerosis. Mult Scler Relat Disord. 2019 Feb;28:221-225. doi: 10.1016/j.msard.2019.01.002. Epub 2019 Jan 3. PMID 30623861
- [Background] Mazhari A. Multiple Sclerosis-Related Pain Syndromes: An Imaging Update. Curr Pain Headache Rep. 2016 Dec;20(12):63. doi: 10.1007/s11916-016-0594-4. PMID 27864731
- [Background] Fallata A, Salter A, Tyry T, Cutter GR, Marrie RA. Trigeminal Neuralgia Commonly Precedes the Diagnosis of Multiple Sclerosis. Int J MS Care. 2017 Sep-Oct;19(5):240-246. doi: 10.7224/1537-2073.2016-065. PMID 29070964
- [Background] Danesh-Sani SA, Rahimdoost A, Soltani M, Ghiyasi M, Haghdoost N, Sabzali-Zanjankhah S. Clinical assessment of orofacial manifestations in 500 patients with multiple sclerosis. J Oral Maxillofac Surg. 2013 Feb;71(2):290-4. doi: 10.1016/j.joms.2012.05.008. Epub 2012 Jun 27. PMID 22742955
- [Background] Kister I, Caminero AB, Monteith TS, Soliman A, Bacon TE, Bacon JH, Kalina JT, Inglese M, Herbert J, Lipton RB. Migraine is comorbid with multiple sclerosis and associated with a more symptomatic MS course. J Headache Pain. 2010 Oct;11(5):417-25. doi: 10.1007/s10194-010-0237-9. Epub 2010 Jul 13. PMID 20625916
- [Background] Zhang GQ, Meng Y. Oral and craniofacial manifestations of multiple sclerosis: implications for the oral health care provider. Eur Rev Med Pharmacol Sci. 2015 Dec;19(23):4610-20. PMID 26698259
- [Background] Foley PL, Vesterinen HM, Laird BJ, Sena ES, Colvin LA, Chandran S, MacLeod MR, Fallon MT. Prevalence and natural history of pain in adults with multiple sclerosis: systematic review and meta-analysis. Pain. 2013 May;154(5):632-642. doi: 10.1016/j.pain.2012.12.002. Epub 2012 Dec 14. PMID 23318126
- [Background] Solaro C, Brichetto G, Amato MP, Cocco E, Colombo B, D'Aleo G, Gasperini C, Ghezzi A, Martinelli V, Milanese C, Patti F, Trojano M, Verdun E, Mancardi GL; PaIMS Study Group. The prevalence of pain in multiple sclerosis: a multicenter cross-sectional study. Neurology. 2004 Sep 14;63(5):919-21. doi: 10.1212/01.wnl.0000137047.85868.d6. PMID 15365151
- [Background] Hadjimichael O, Kerns RD, Rizzo MA, Cutter G, Vollmer T. Persistent pain and uncomfortable sensations in persons with multiple sclerosis. Pain. 2007 Jan;127(1-2):35-41. doi: 10.1016/j.pain.2006.07.015. Epub 2006 Sep 1. PMID 16949751
- [Background] Labuz-Roszak B, Niewiadomska E, Kubicka-Baczyk K, Skrzypek M, Tyrpien-Golder K, Majewska A, Matejczyk A, Dobrakowski P, Pierzchala K. Prevalence of pain in patients with multiple sclerosis and its association with anxiety, depressive symptoms and quality of life. Psychiatr Pol. 2019 Apr 30;53(2):475-486. doi: 10.12740/PP/94469. Epub 2019 Apr 30. English, Polish. PMID 31317971